CLINICAL TRIAL: NCT05238727
Title: Effect of Volume Increase Compared to Supplemental 4% Articaine Buccal Infiltration on Mepivacaine Inferior Alveolar Nerve Block Success in Cases With Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: Volume Increase Versus Supplemental 4% Articaine Buccal Infiltration on Mepivacaine Inferior Alveolar Nerve Block Success
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Anwar Mohammed El Said Sleem, Ms, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CU-ENDO-2-2-2022.
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Symptomatic Irreversible Pulpitis
MeSH Terms: interventions — Mepivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1.8 ml mepivacaine IANB (Active Comparator)
  Interventions: Drug: 1.8 ml mepivacaine hydrochloride
- 3.6 ml mepivacaine IANB (Experimental)
  Interventions: Drug: 3.6 ml mepivacaine hydrochloride
- 1.8 ml mepivacaine IANB plus 1.8 ml articaine BI (Experimental)
  Interventions: Drug: 1.8 ml mepivacaine hydrochloride IANB plus 1.8 ml articaine hydrochloride BI

INTERVENTIONS:
Drug: 1.8 ml mepivacaine hydrochloride — 1.8 ml mepivacaine IANB
  Arms: 1.8 ml mepivacaine IANB
Drug: 3.6 ml mepivacaine hydrochloride — 3.6 ml mepivacaine IANB
  Arms: 3.6 ml mepivacaine IANB
Drug: 1.8 ml mepivacaine hydrochloride IANB plus 1.8 ml articaine hydrochloride BI — 1.8 ml mepivacaine IANB plus 1.8 ml articaine BI
  Arms: 1.8 ml mepivacaine IANB plus 1.8 ml articaine BI

SUMMARY:
To assess the anesthetic success of inferior alveolar nerve block (IANB), intraoperative pain intensity and need for supplemental anesthesia on administration of 1.8ml or 3.6ml 2% mepivacaine IANB, or 1.8ml 2% mepivacaine IANB plus 1.8ml 4% articaine buccal infiltration (BI) in mandibular molars with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
Patients with moderate-to-severe preoperative pain related to mandibular molars with symptomatic irreversible pulpitis will be included. Patients receive 1.8 ml, 3.6 ml 2% mepivacaine IANB, or 1.8ml 2% mepivacaine IANB plus 1.8ml 4% articaine BI. Anesthetic success of inferior alveolar nerve block, intraoperative pain intensity and need for supplemental anesthesia will be assessed during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in good health (ASA Class I, II).
2. Age between 18-60 years old.
3. Males or females.
4. Mandibular molar teeth diagnosed with symptomatic irreversible pulpitis.
5. Patients who can understand NRS scale and sign the informed consent.

Exclusion Criteria:

1. Patients who had used any type of analgesic medication during the preceding 8 hours before the treatment.
2. Pregnant or nursing females.
3. Patients with a contraindication for the use of mepivacaine, articaine or any used drug or material.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Anesthetic success | During the treatment
  Will be recorded by 11-point numerical rating scale (NRS) consisting of numbers from 0 through 10. 0: reading represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain". Success will be defined as no to mild pain.

SECONDARY OUTCOMES:
Intraoperative pain | During the treatment
  Will be recorded by 11-point numerical rating scale (NRS) consisting of numbers from 0 through 10. 0: reading represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain".
Need for supplemental anesthesia | During the treatment
  Whether the patient requires supplemental anesthesia or not

REFERENCES:
- [Background] Abazarpoor R, Parirokh M, Nakhaee N, Abbott PV. A Comparison of Different Volumes of Articaine for Inferior Alveolar Nerve Block for Molar Teeth with Symptomatic Irreversible Pulpitis. J Endod. 2015 Sep;41(9):1408-11. doi: 10.1016/j.joen.2015.05.015. Epub 2015 Jul 3. PMID 26149210
- [Background] Aggarwal V, Singla M, Miglani S, Kohli S, Singh S. Comparative evaluation of 1.8 mL and 3.6 mL of 2% lidocaine with 1:200,000 epinephrine for inferior alveolar nerve block in patients with irreversible pulpitis: a prospective, randomized single-blind study. J Endod. 2012 Jun;38(6):753-6. doi: 10.1016/j.joen.2012.02.003. Epub 2012 Mar 3. PMID 22595107
- [Background] Parirokh M, Satvati SA, Sharifi R, Rekabi AR, Gorjestani H, Nakhaee N, Abbott PV. Efficacy of combining a buccal infiltration with an inferior alveolar nerve block for mandibular molars with irreversible pulpitis. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Mar;109(3):468-73. doi: 10.1016/j.tripleo.2009.11.016. PMID 20219602